CLINICAL TRIAL: NCT02925013
Title: Maternal Dietary Lipids and Omega 3 Essential Fatty Acids Profile in Pregnant Women at Term and Their Fetuses
Acronym: OM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9649-12
Record Dates: First submitted 2016-09-27; First posted 2016-10-05 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Lipid Profile in Pregnancy
Keywords: Omega 3; Lipids; Pregnancy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Pregnant women at delivery
  Interventions: Procedure: Blood sampling; Other: Dietary- Normal western diet
- Control group (Other): Women in fertility age not pregnant
  Interventions: Procedure: Blood sampling; Other: Dietary- Normal western diet

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling for lipid profile
Other: Dietary- Normal western diet — Normal western diet

SUMMARY:
This study aims to investigate the omega 3 lipid profile in pregnant women at term and their fetuses compared to non pregnant women , in normal western diet adding no supplementation

DETAILED DESCRIPTION:
DHA (Docosahexaenoic Acid ) is a long chain omega-3 fatty acid important for brain and eye development and function throughout life. It also supports heart health. DHA is the most abundant omega-3 in the brain and retina and is naturally found in breast milk. EPA (Eicosapentaenoic Acid ) is a long-chain omega-3 fatty acid important for overall health. However, unlike DHA, the body does not store EPA in significant quantities in the brain or retina (DHA is found in every cell throughout the body, EPA is not). These Omega 3 fatty acids are considered essential due to the inability of the human body to create them and the need to consume them from nutritional source. Food that is considered rich in omega 3 fatty acids are fat fish and green vegetables. Omega-3 fatty acids are "good fats," and are among the most important nutrients lacking in Western diets today. The average person in developed countries consumes less than 100 mg of DHA daily. With increasing awareness of the importance of DHA, many people realize that they need to make a change to their diet by adding DHA-rich foods or supplements.

Alpha Linolenic Acid (ALA) is a shorter-chain omega-3 that serves as a source of energy and as a building block for long-chain omega-3 fatty acids (DHA and EPA). This precursor for omega 3 fatty acid is abundant in falx seeds. The mother and the fetus has the metabolic mechanism that enables them to transform ALA into EPA,DHA endogenously.

Women during pregnancy are predisposed to a reduction in unsaturated long chain fatty acid (polyunsaturated Fatty Acid = PUFA) from the omega 3 group . Lately, a new hypothesis claiming that a reduced level of this essential acids expose the fetus later in his adult life to a spectrum of metabolic and cardiovascular disease. New publication on animal models showed higher rates of obesity, insulin resistance diabetes and cardiovascular damage on mice exposed short chain fatty acids compared to those treated with enriched ALA diet supplementation. Different nutritional and gynecological health organization around the world including the FDA, recommend incorporating omega 3 fatty acids supplementation to daily diet and specifically in pregnant women in order to raise their blood levels for the developing fetus. However, normal fatty acid profile of the omega 3 group in mother and fetus haven't been described yet . Furthermore, the total effect and future benefit to fetus haven't been thoroughly studied and is based mainly on presumptions.

The aim of this study is to learn the typical omega 3 fatty acid profile at women near delivery and their fetuses and to compare it to women in productive years that are not pregnant.

Study methods:

Women close to term visiting the obstetrical triage and fitting inclusion criteria will be offered to participate in the study. Demographic medical and obstetrical information will be collected from medical files after giving signed informed consent .

Blood sample ( one blood tube that will include 5 cc of blood ) will be taken while insertion of intravenous line in the delivery room, and another blood sample will be taken from the umbilical vein after delivery and separation of the fetus from the umbilical cord.

Women for control group - healthy non pregnant women in fertility years, will be recruited from the gynecological clinic . Similarly to the study group, one of the study researchers will collect one tube for blood sampling ( equal to 5 cc of blood ).

All samples will be sent for profile analysis of omega 3 fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in labor( above 34 weeks of gestation )
* Age:18-42

Exclusion Criteria:

* taking any kind of dietary supplementation
* hyperlipidemia / hypercholesterolemia

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Omega 3 lipid profile in pregnant women at term | through study completion, an average of 1year
Omega 3 lipid profile in umbilical vein | through study completion, an average of 1year
Omega 3 lipid profile in women in fertility age | through study completion, an average of 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Mennitti LV, Oliveira JL, Morais CA, Estadella D, Oyama LM, Oller do Nascimento CM, Pisani LP. Type of fatty acids in maternal diets during pregnancy and/or lactation and metabolic consequences of the offspring. J Nutr Biochem. 2015 Feb;26(2):99-111. doi: 10.1016/j.jnutbio.2014.10.001. Epub 2014 Oct 12. PMID 25459884
- [Background] Leikin-Frenkel AI. Is there A Role for Alpha-Linolenic Acid in the Fetal Programming of Health? J Clin Med. 2016 Mar 23;5(4):40. doi: 10.3390/jcm5040040. PMID 27023621
- [Background] Barker DJ. Fetal origins of coronary heart disease. Br Heart J. 1993 Mar;69(3):195-6. doi: 10.1136/hrt.69.3.195. No abstract available. PMID 8461215
- [Background] Hollander KS, Tempel Brami C, Konikoff FM, Fainaru M, Leikin-Frenkel A. Dietary enrichment with alpha-linolenic acid during pregnancy attenuates insulin resistance in adult offspring in mice. Arch Physiol Biochem. 2014 Jul;120(3):99-111. doi: 10.3109/13813455.2014.940352. Epub 2014 Jul 17. PMID 25030769
- [Background] Shomonov-Wagner L, Raz A, Leikin-Frenkel A. Alpha linolenic acid in maternal diet halts the lipid disarray due to saturated fatty acids in the liver of mice offspring at weaning. Lipids Health Dis. 2015 Feb 26;14:14. doi: 10.1186/s12944-015-0012-7. PMID 25889505
- [Background] Leikin-Frenkel A, Shomonov-Wagner L, Juknat A, Pasmanik-Chor M. Maternal Diet Enriched with alpha-Linolenic or Saturated Fatty Acids Differentially Regulates Gene Expression in the Liver of Mouse Offspring. J Nutrigenet Nutrigenomics. 2015;8(4-6):185-94. doi: 10.1159/000442945. Epub 2016 Jan 21. PMID 26788914
- [Background] Kabaran S, Besler HT. Do fatty acids affect fetal programming? J Health Popul Nutr. 2015 Aug 13;33:14. doi: 10.1186/s41043-015-0018-9. PMID 26825664